CLINICAL TRIAL: NCT01280682
Title: Immune Intervention With Anti-CD20 Monoclonal Antibody to Preserve Beta Cell Function in Early Onset Type 1 Diabetes
Brief Title: Immune Intervention With Rituximab to Preserve Beta Cell Function in Early Onset Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yang Tao (Other)
Responsible Party: Sponsor-Investigator, Yang Tao, Department of Endocrinology & Metabolism, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-SR-021
Record Dates: First submitted 2010-07-29; First posted 2011-01-21 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; age; course of disease; autoantibodies; C-peptide levels
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rituximab (Experimental): patients who had newly diagnosed type 1 diabetes are assigned to receive infusions of rituximab of 125mg/m^2 day1 day8 day15 day22 repeat after six months (only day1 and day8) besides insulin
  Interventions: Drug: rituximab
- parallel control (No Intervention): patients who had newly diagnosed type 1 diabetes only use insulin

INTERVENTIONS:
Drug: rituximab — anti-CD20 monoclonal antibody 125mg/m^2 day1 day8 day15 day22 repeat after six months (only day1 and day8)
  Other Names: anti-CD20 monoclonal antibody
  Arms: rituximab

SUMMARY:
Transient elimination of B lymphocytes with anti-CD20 monoclonal antibody would decrease immune-mediated destruction of beta cells and result in preserved beta-cell function in patients with type 1 diabetes of recent onset.

DETAILED DESCRIPTION:
Although the presence of autoantibodies is a diagnostic criterion, the immunopathogenesis of beta-cell destruction in type 1 diabetes is typically associated with T-lymphocyte autoimmunity.

Many T-lymphocyte-mediated diseases include a B-lymphocyte component. B lymphocytes can play a crucial role as antigen-presenting cells, expressing high levels of class II major-histocompatibility-complex antigens and generating cryptic peptides to which T lymphocytes are not tolerant.

B lymphocytes can be selectively depleted with the anti-CD20 monoclonal antibody. We will test the hypothesis that transient elimination of B lymphocytes with anti-CD20 monoclonal antibody would decrease immune-mediated destruction of beta cells and result in preserved beta-cell function in patients with type 1 diabetes of recent onset.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 1 diabetes
* The age of subjects between 8 and 70 years old
* Course of disease within 12 months
* Presence of at least one type of detectable islet autoantibody [zinc transporter 8 antibody(ZnT8A),glutamic acid decarboxylase antibody(GADA),protein tyrosine phosphatase-2 antibody(IA-2A),insulin autoantibody(IAA)]
* Fasting C-peptide levels of at least 0.2 pmol/mL

Exclusion Criteria:

* Confirmed diagnosis of type 2 diabetes
* Severe chronic or acute complications of diabetes
* Severe infection or damage to the immune response
* Presence of chronic latent infection in vivo
* Viral hepatitis B patients whose hepatitis B virus(HBV)DNA > log10^5
* Liver and kidney dysfunction, alanine aminotransferase(ALT), aspartate aminotransferase(AST), and creatinine more than 2 times the upper limit of normal
* Hypotension, systolic blood pressure(SBP) ≤ 90mmHg, diastolic blood pressure(DBP) ≤ 60mmHg
* Patients with rheumatoid arthritis
* Allergic to any component of this drug
* Pregnancy, breast-feeding women
* Use of other immunosuppressive agents 3 months before selected

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, MD/PhD, Principal Investigator — First Affiliated Hospital, Nanjing Medical University, China
Locations (1):
- First Affiliated Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Su Z, Ma C, Zhao R, Jiang Y, Cai Y, Yong G, Yang T, Xu X. Heterogeneity of circulating CXCR5-PD-1hiTph cells in patients of type 2 and type 1 diabetes in Chinese population. Acta Diabetol. 2023 Jun;60(6):767-776. doi: 10.1007/s00592-023-02055-6. Epub 2023 Mar 6. PMID 36879107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients who had newly diagnosed type 1 diabetes
Pre-assignment Details: patients whose C-peptide were too low
Groups:
- Paralelle Control Group: patients who had newly diagnosed type 1 diabetes only used insulin.
- Rituximab Group: besides insulin, patients who had newly diagnosed type 1 diabetes are assigned to receive infusions of rituximab (125 mg per square meter of body-surface area) in a solution (pH 6.5) with 9 mg of sodium chloride per milliliter on days 1, 8, 15, and 22 of the study.
Period: Overall Study
Arm/Group | Paralelle Control Group | Rituximab Group
Started | 30 | 90
Completed | 30 | 77
Not Completed | 0 | 13
Not completed — Lost to Follow-up | 0 | 6
Not completed — Withdrawal by Subject | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Rituximab: patients who had newly diagnosed type 1 diabetes are assigned to receive infusions of rituximab besides insulin
- Parallel Control: patients who had newly diagnosed type 1 diabetes only used insulin
- Total: Total of all reporting groups
Arm/Group | Rituximab | Parallel Control | Total
Number analyzed (Participants) | 77 | 30 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 17 | 68
  Between 18 and 65 years | 26 | 13 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.81 (8.76) | 20.08 (7.40) | 18.27 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 14 | 46
  Male | 45 | 16 | 61
Region of Enrollment [Number; unit: participants]
  China | 77 | 30 | 107

OUTCOME MEASURES:

1. Primary Outcome: Change of 3-hour Mean Area Under the Curve (AUC) of C-peptide
Description: Change of 3-hour mean area under the curve (AUC) of C-peptide at 6 months from baseline. AUC was calculated from C-peptide timing measurements during the 3-hour mixed meal tolerance test with the trapezoidal rule. The mean AUC for C-peptide is equal to the calculated AUC divided by the 3 h interval (i.e., AUC/180). All mean C-peptide AUC data were transformed as log (mean AUC) for analysis.
Time Frame: 6 months after participants completed the injection
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Rituximab | Parallel Control
Number analyzed (Participants) | 77 | 30
pmol/L | -0.01 (0.03) | -0.35 (0.05)

2. Secondary Outcome: Change of Fasting C-peptide
Description: The change of fasting level of C-peptide during the 3-hour of a mixed meal tolerance test at 6 months from baseline. All fasting C-peptide data were transformed as log (fasting C-peptide) for analysis.
Time Frame: 6 months after participants completed the injection
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Rituximab | Parallel Control
Number analyzed (Participants) | 77 | 30
pmol/L | -0.03 (0.04) | -0.34 (0.07)

3. Secondary Outcome: Change of Peak C-peptide
Description: The change of peak level of C-peptide during the 3-hour of a mixed meal tolerance test at 6 months from baseline. All peak C-peptide data were transformed as log (peak C-peptide) for analysis.
Time Frame: 6 months after participants completed the injection
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Rituximab | Parallel Control
Number analyzed (Participants) | 77 | 30
pmol/L | -0.01 (0.03) | -0.29 (0.06)

4. Secondary Outcome: HbA1c Levels
Description: Glycated hemoglobin (HbA1c) levels (%)
Time Frame: 6 months after participants completed the injection
Measure: Mean (95% Confidence Interval); unit: percentage of hemoglobin
Arm/Group | Rituximab | Parallel Control
Number analyzed (Participants) | 77 | 30
percentage of hemoglobin | 6.84 [6.50 to 7.17] | 9.35 [7.54 to 11.15]

ADVERSE EVENTS:
Arm/Group | Rituximab | Parallel Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/30
Other Adverse Events (participants affected / at risk) | 44/77 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=77) | Parallel Control (N=30)
Fever (General disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Cardiac disorders) | 2 | 0
Hypertension (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 15 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0
Other AE (General disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes